CLINICAL TRIAL: NCT00493701
Title: ADAPT-The Adaptation to High Fat Diets
Brief Title: "ADAPT" The Adaptation to High Fat Diets Extention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PBRC 21041
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle (Other): Measurement of body weight in a fown with light undercloting (30 minutes) and height.
  Interventions: Behavioral: High Fat Diet
- DEXA Scanner (Other): Low-dose X0rays to determine the amount of fat, bone and muscle in your body.
  Interventions: Behavioral: Low Fat Diet

INTERVENTIONS:
Behavioral: High Fat Diet — Daily eating
  Other Names: Measurements will be collected to help with gathering data.
  Arms: Lifestyle
Behavioral: Low Fat Diet — Life style eating habits
  Other Names: Questionnairs of food frequency
  Arms: DEXA Scanner

SUMMARY:
This study is designed to predict weight gain overtime after a high fat diet.

DETAILED DESCRIPTION:
In the past 3 years we have identified a "thrifty-phenotype" characterized in lean men by an inability to adapt rapidly to a high fat diet and associated with a low maximal VO2 and high fasting insulin. We hypothesize that the individuals with the "thrifty phenotype" are at higher risk for becoming obese, and that exercise may be effective in overcoming this problem.

Several questions remain to be answered regarding the "thrifty" phenotype. First, given the large interindividual differences, how can we identify those at the highest risk? What are the distinguishing biochemical, endocrine and environmental characteristics of individuals that store fat when exposed to high fat diets? This is important because if these individuals can be easily identified, then dietary interventions can be targeted to this "at-risk" population.

Second, what is different about the individual with the "thrifty phenotype"? Are there cellular pathways that are dysregulated in the skeletal muscle of these individuals when compared to controls? Is the defect intrinsic, i.e. a diminished ability to conserve glucose and oxidize fat in skeletal muscle or alternately, is the phenotype due to environmental, and dietary factors such as inactivity and energy excess?

To answer these questions, we have planned a three-year project that aims to:

* Characterize the biochemical, endocrine, anthropometric and environmental characteristics of individuals with the "thrifty" phenotype.
* Identify the signaling pathways in skeletal muscle that are dysregulated in individuals with the "thrifty" phenotype through mRNA expression profiling in skeletal tissue.
* Determine the role of environmental factors such as inactivity and caloric intake vs. intrinsic (genetic) factors in the "thrifty" phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Both genders and all races will be invited to participate
* Women will be asked to participate in the follicular phase of the menstrual cycle as determined by menstrual history and a negative pregnancy test will be recorded prior to participation
* BMI > 19 and < 35
* Age 18-30 Exclusion Criteria
* Smokers
* Unwilling or unable to abstain from alcohol consumption and caffeine consumption prior to testing and laboratory
* Significant renal, hepatic, endocrine, pulmonary, cardiac or hematological disease
* Pregnancy
* Corticosteroid use in previous two months
* Chronic use of anti-diabetic, anti-hypertensive, or other medications known to affect fat metabolism
* Use of Depo-Provera, hormone implants or estrogen replacement therapy
* Irregular menstrual cycles
* Post-menopausal women
* Weight gain or loss of > 3kg in the last 6 months

For the MRI, the following exclusion criteria apply:

* Individuals who have a heart pacemaker, defibrillator, or non-removable hearing aid
* Individuals with any clips or metal plates in their head
* Individuals who have any artificial limbs or prosthetic devices
* Individuals who were ever injured by a metallic foreign body which was not removed
* Individuals, who wear braces on their teeth, have non-removable false teeth, or removable bridgework

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Characteristics of Individuals | 4 days of high fat diet
  Characterize the biochemical, endocrine, anthropometric and environmental characteristics of individuals with the "thrifty" phenotype.

SECONDARY OUTCOMES:
Identify the Signaling Pathways | 4 days after high fat diet
  Identify the signaling pathways in skeletal muscle that are dysregulated in individuals with the "thrifty" phenotype through mRNA expression profiling in skeletal tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151
- [Derived] Pasarica M, Xie H, Hymel D, Bray G, Greenway F, Ravussin E, Smith SR. Lower total adipocyte number but no evidence for small adipocyte depletion in patients with type 2 diabetes. Diabetes Care. 2009 May;32(5):900-2. doi: 10.2337/dc08-2240. Epub 2009 Feb 19. PMID 19228873